CLINICAL TRIAL: NCT02876432
Title: Evaluating Acupuncture in the Treatment of Low Back Pain in Athletes and the Relationship With the Catecholaminergic Pathway
Brief Title: Evaluating Acupuncture Relationship With the Catecholaminergic Pathway
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autónoma Benito Juárez de Oaxaca (Other)
Responsible Party: Principal Investigator, Rafael Torres Rosas, Full Time Professor Researcher, Universidad Autónoma Benito Juárez de Oaxaca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: PEL0011FO
Record Dates: First submitted 2016-08-16; First posted 2016-08-23 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Electroacupuncture; Diclofenac

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Device: Electroacupuncture (Experimental): The acupuncture points selected were ST36, BL25, GB30, BL40, GB34 the needles were inserted into acupoints and the depth of needle insertion depended of the acupoints selected to achieve Deqi sensation, which is characterized as a numb, heavy, sore and/or distending sensation.
  Electrical stimulation was delivered at 4 Hz. The stimulator (ITO EST-160) was then switched on, and the intensity was gradually increased to reach a strong but comfortable level the sensation of EA which is characterized for numbness, tingling and a light muscle cramp. For 15 minutes
  Interventions: Device: Electroacupuncture; Other: Sham electroacupuncture
- Device: Sham Electroacupuncture (Sham Comparator): In sham electroacupuncture (Sham) the investigators use 1.0 cm outside point of the real electroacupuncture, the depth of needle insertion was superficial to avoid Deqi sensation, the cables wasn't connected to the electro stimulator and was then switched on for 15 minutes. The participants were threaded separately to avoid sharing experiences about the electroacupuncture sessions
  Interventions: Device: Electroacupuncture; Other: Sham electroacupuncture
- Drug: Diclofenac sodium (Active Comparator): 100 mg Diclofenac sodium was administrated orally every 12 hours for 5 days.
  Interventions: Drug: Diclofenac sodium

INTERVENTIONS:
Device: Electroacupuncture — The acupuncture points selected were ST36, BL25, GB30, BL40, GB34 the needles were inserted into acupoints and the depth of needle insertion depended of the acupoints selected to achieve Deqi sensation, which is characterized as a numb, heavy, sore and/or distending sensation.
  Electrical stimulation was delivered at 4 Hz. The stimulator (ITO EST-160) was then switched on, and the intensity was gradually increased to reach a strong but comfortable level the sensation of EA which is characterized for numbness, tingling and a light muscle cramp. For 15 minutes
  Arms: Device: Electroacupuncture; Device: Sham Electroacupuncture
Drug: Diclofenac sodium — 100 mg Diclofenac sodium was administrated orally every 12 hours for 5 days.
  Arms: Drug: Diclofenac sodium
Other: Sham electroacupuncture — The investigators use 1.0 cm outside point of the real electroacupuncture, the depth of needle insertion was superficial to avoid Deqi sensation, the cables wasn't connected to the electro stimulator and was then switched on for 15 minutes. The participants were threaded separately to avoid sharing experiences about the electroacupuncture sessions
  Arms: Device: Electroacupuncture; Device: Sham Electroacupuncture

SUMMARY:
Activation of the sympathetic nervous system attenuates inflammation via catecholamines, recent advances in electroacupuncture allow activating critical neuronal networks with the release of catecholamines the aim of this research was to evaluate de effect of electroacupuncture in the activation of sympathetic nervous system and the control of low back pain in athletes

DETAILED DESCRIPTION:
Activation of the sympathetic nervous system attenuates inflammation via activation of β2-adrenoreceptors by catecholamines, Electrical stimulation of vagus nerve limits the inflammatory response in several animal models of inflammatory diseases, In addition, voluntary activation of the sympathetic nervous system by meditation, training or breathing techniques limits production of proinflammatory cytokines in vivo during experimental endotoxemia in healthy human volunteers.

Currently there are therapies that effectively antagonize proinflammatory cytokines and control pain, as non-steroidal anti-inflammatory drugs and opioid analgesics, but had serious side effects if used chronically. Therefore, alternative therapies as electroacupuncture, which may limit inflammatory cytokine production more physiologically, are warranted. The aim of this study was to evaluate de effect of electroacupuncture used for attenuation of low back pain in the activation of sympathetic nervous system and leukocyte inflammatory potential.

ELIGIBILITY:
Inclusion Criteria:

(Controls)

* Healthy
* Non Smokers
* Athletes

(Cases)

* Acute Low Back Pain (less than 1 month)
* Athletes
* Non Smokers

Exclusion Criteria:

* Sciatic Pain
* Smokers
* Chronic Low Back Pain

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | before Electroacupuncture Time "0"
  in a horizontal line, 100 mm in length, anchored by word descriptors at each end. The patient marks on the line the point that they feel represents their perception of their current state.
  The VAS score is determined by measuring in millimetres from the left hand end of the line to the point that the patient marks
Levels of catecholamines in serum | five minutes before Electroacupuncture
  Blood was collected into chilled heparin tubes serum catecholamines were determined by ELISA (Rocky Mountain Diagnostics, Colorado Springs, CO)

SECONDARY OUTCOMES:
Levels of catecholamines in serum | five minutes after Electroacupuncture
  Blood was collected into chilled heparin tubes serum catecholamines were determined by ELISA (Rocky Mountain Diagnostics, Colorado Springs, CO)
Visual analogue scale | Five days after Electroacupuncture
  in a horizontal line, 100 mm in length, anchored by word descriptors at each end. The patient marks on the line the point that they feel represents their perception of their current state.
  The VAS score is determined by measuring in millimetres from the left hand end of the line to the point that the patient marks

CONTACTS AND LOCATIONS:
Overall Officials: Lourdes Arriaga Pizano, MD PhD, Study Director — IMSS

IPD SHARING:
Plan to Share IPD: No